CLINICAL TRIAL: NCT05606627
Title: A Study on Correlation Between Antibiotics Resistance and Incidence of Sepsis in Community Acquired Pneumonia in RICU Patients, Assiut University Hospital.
Brief Title: Correlation Between Antibiotic Resistance and Incidence of Sepsis in Community Acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdelrhman Kotb Said, Resident doctor, Assiut University
Other Study IDs: Community Acquired pneumonia
Record Dates: First submitted 2022-10-22; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Community-acquired Pneumonia; Antibiotic Resistance; Sepsis
MeSH Terms: conditions — Community-Acquired Pneumonia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Correlation between antibiotic resistance and incidence of sepsis in community acquired pneumonia in RICU patients.

DETAILED DESCRIPTION:
Adult community-acquired pneumonia (CAP) is a leading cause of morbidity, often needing hospitalization, and an important cause of mortality, especially in severe cases with sepsis or requiring assisted ventilation[1]. Typical bacterial pathogens that cause CAP include Streptococcus pneumoniae, Haemophilus influenzae, and Moraxella catarrhalis[2].

Clinical diagnosis is based on a group of signs and symptoms related to lower respiratory tract infection with presence of fever >38ºC (>100ºF), cough, muco purulent sputum, pleuritic chest pain, dyspnoea, and new focal chest signs on examination such as crackles or bronchial breathing[3]. There are numerous tools such as the Pneumonia Severity Index (PSI) and the CURB-65 (confusion, urea, respiratory rate, blood pressure and age ≥65) score to identify and evaluate indication of ICU admission [4].Sever CAP patients may develop signs and symptoms of systemic inflammatory response syndrome (SIRS).

Systemic inflammatory response syndrome (SIRS) is an exaggerated defense response of the body to a noxious stressor (infection, trauma, surgery, acute inflammation, ischemia or reperfusion, or malignancy, to name a few) to localize and then eliminate the endogenous or exogenous source of the insult[8]. Criteria of SIRS heart rate greater than 90, respiratory rate greater than 20, temperature greater or equal to 38 ⁰ C or less than 36⁰ C, altered mental state and one of the following risk factors should be considered at risk of sepsis:Looks unwell, Age greater than 65 years, Recent surgery, Immunocompromised (AIDS, chemotherapy, neutropenia, transplant, chronic steroids), Chronic illness (diabetes, renal failure, hepatic failure, cancer, alcoholism, IV drug use )[8]Table [1] .When SIRS caused by infectious cause (Bacteria, Vairus, Fungi,…etc) and associated with multiorgan dysfunction is defined as sepsis.

Sepsis and septic shock are medical emergencies, and studies recommend that treatment and resuscitation begin immediately[8]. Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. Septic shock is a life-threatening condition that happens when blood pressure drops to a dangerously low level after an infection[9]. Septic shock is defined by persisting hypotension requiring vasopressors to maintain a mean arterial pressure of 65 mm Hg or higher and a serum lactate level greater than 2 mmol/L (18 mg/dL) despite adequate volume resuscitation.

Recent studies suggests that there is a relationship between antibiotic resistance and the incidence of sepsis in community-acquired bacterial pneumonia and considered it one of the most significant health complications that can result from antimicrobial resistance.As more germs become resistant to antimicrobial medicines used to treat infection, more people are at risk for developing sepsis.

According to WHO, widespread use and abuse of antibiotics have led to the rapid emergence and spread of antimicrobial resistance globally, and empirical management of CAP is rendered difficult (for a choice of drug, as most drugs are ineffective) by this phenomenon[5]. Antimicrobial Resistance (AMR) occurs when bacteria, viruses, fungi and parasites change over time and no longer respond to medic medicines making infections harder to treat and increasing the risk of disease spread, severe illness and death[6]. Four major AMR risk factor domains were identified: (1) sociodemographic factors (includes migrant status, low income and urban residence), (2) patient clinical information (includes disease status and certain laboratory results), (3) admission to healthcare settings (includes length of hospitalisation and performance of invasive procedures) and (4) drug exposure (includes current or prior antibiotic therapy)[7].

So , The primary end point of this study is assessment the correlation between drug resistance and incidence of sepsis and the secondry end point is improving mortality and morbidity of patients with sever CAP in ICU.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients above 18 yrs. old. 2. Patients with sever community acquired bacterial pneumonia confirmed by clinical symptoms (CURB-65 scores >= 4) and culture.

3.Informed consent to participate in the study is provided.

Exclusion Criteria:

- 1. Patients below 18 yrs. old. 2. Patient don't meet the criteria of community acquired bacterial pneumonia (viral, fungal, chemical,…etc.).

3. Patients with comorbid respiratory diseases. 4. Patients with Hospital acquired pneumonia. 5. Patients receiving empirical antibiotics. 6. Patients receiving anti-TB drugs, systemic steroids or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to RICU with sever community acquired pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
1.Define antibiotic resistant organisms 2.Assess correlation between antibiotic resistance and incidence of sepsis in CAP patiants 3. Assess incidence of sepsis in CAP patiants using SOFA score. | October 2022/ April 2024

SECONDARY OUTCOMES:
1.Decrease MDR phenomenon 2.improving mortality and morbidity of patients with sever CAP in ICU. | October 2022/April 2024